CLINICAL TRIAL: NCT03912506
Title: Severe Leptospirosis in Non-tropical Areas: a Nationwide, Multicentre, Retrospective Study in French ICUs
Brief Title: Severe Leptospirosis in Non-tropical Areas
Acronym: LEPTOREA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LEPTOREA
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Leptospirosis; Intensive Care Unit; Epidemiology; Alveolar Hemorrhage
MeSH Terms: conditions — Leptospirosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient admitted in the ICU for leptospirosis: Patient admitted in the ICU for leptospirosis None intervention was performed according to retrospective design

SUMMARY:
Leptospirosis is a worldwide zoonosis. The mortality of the disease is between 3,6% to 13%, and up to 48% for the severe leptospirosis.

Only few studies exist on severe leptospirosis and none major multicentre on leptospirosis in intensive care units in Europe. The investigators conduct a retrospective multi centric study in metropolitan France in order to identify the characteristic, the treatments and the prognostic factors associated with mortality of sever leptospirosis.

DETAILED DESCRIPTION:
Leptospirosis is a worldwide zoonosis. The infection is acquired through contact with animal urine on contaminated soil. It is an important remerging infectious disease because of its increasing incidence. Leptospirosis is most common in tropical and rural settings but its incidence has been constantly increasing for the past ten years in Metropolitan France. Most of the cases are asymptomatic or sparsely symptomatic, but some patients develop severe leptospirosis (6% to 59%), requiring hospitalisation in intensive care units. The mortality of the disease is between 3,6% to 13%, and up to 48% for the severe leptospirosis.

Only few studies exist on severe leptospirosis and none major multicentre on leptospirosis in intensive care units in Europe. Therefore, the investigators have decided to carry out this studies. The investigators conduct a retrospective multi centric study in metropolitan France in order to identify the characteristic, the treatments and the prognostic factors associated with mortality of sever leptospirosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in ICU
* Leptospirosis confirmed with one laboratory test (MAT, ELISA, PCR, direct examination)

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in participating ICUs between January 2012 and September 2016 and diagnosed having leptospirosis were included in the study. Patients were identified by searching code A27 in the hospitals databases for International Statistical Classification of Diseases and Related Health Problems, 10th revision
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Mortality at ICU discharge | ICU discharge (usually 5 days)
  Mortality was evaluated at ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jean Reignier, MD, PhD, Study Director — Nantes University Hospital
Locations (36):
- France (36):
  - CHU Amiens-Picardie, Amiens
  - CHU Angers, Angers
  - CH Angoulème, Angoulême
  - CH Annecy, Annecy
  - CH Avignon, Avignon
  - hopital saint Leon, CH de la Cote Basque, Bayonne
  - CHU Besançon, Besançon
  - CH Fleyriat, Bourg-en-Bresse
  - CHU de Caen, Caen
  - CH Cahors, Cahors
  - CH Chartres, Chartres
  - CH Cholet, Cholet
  - CHD de la Vendée, La Roche-sur-Yon
  - Hopital Saint Louis, La Rochelle
  - CH Le Mans, Le Mans
  - CH Lens, Lens
  - CHU de Lille, Lille
  - Hopital Edouard Herriot, Hospices civils de Lyon, Lyon
  - GHR MSA, Mulhouse
  - CHRU de Nancy, Nancy
  - CH Niort, Niort
  - CHU Bicetre APHP, Paris
  - CHU Cochin APHP, Paris
  - CHU Henri Mondor, Paris
  - CHU Saint Louis, APHP, Paris
  - CH Périgueux, Périgueux
  - CH René-Dubost, Pontoise
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CH Saint Brieuc, Saint-Brieuc
  - CH Saint Nazaire, Saint-Nazaire
  - CH Saint Malo, St-Malo
  - CHRU Bretonneau, Tours
  - CH Valenciennes, Valenciennes
  - CH Vannes, Vannes
  - Hopital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haake DA, Levett PN. Leptospirosis in humans. Curr Top Microbiol Immunol. 2015;387:65-97. doi: 10.1007/978-3-662-45059-8_5. PMID 25388133
- [Background] Picardeau M. Virulence of the zoonotic agent of leptospirosis: still terra incognita? Nat Rev Microbiol. 2017 May;15(5):297-307. doi: 10.1038/nrmicro.2017.5. Epub 2017 Mar 6. PMID 28260786
- [Background] Delmas B, Jabot J, Chanareille P, Ferdynus C, Allyn J, Allou N, Raffray L, Gauzere BA, Martinet O, Vandroux D. Leptospirosis in ICU: A Retrospective Study of 134 Consecutive Admissions. Crit Care Med. 2018 Jan;46(1):93-99. doi: 10.1097/CCM.0000000000002825. PMID 29116996
- [Background] Costa F, Hagan JE, Calcagno J, Kane M, Torgerson P, Martinez-Silveira MS, Stein C, Abela-Ridder B, Ko AI. Global Morbidity and Mortality of Leptospirosis: A Systematic Review. PLoS Negl Trop Dis. 2015 Sep 17;9(9):e0003898. doi: 10.1371/journal.pntd.0003898. eCollection 2015. PMID 26379143